CLINICAL TRIAL: NCT00627952
Title: Double Blind, Randomized, Parallel Group, Multicentre Study to Evaluate the Effects of Manidipine 20 MG Vs. Amlodipine 10 MG and the Combination of Manidipine 10 MG Plus Delapril 30 MG Vs. Amlodipine 5 MG Plus Delapril 30 MG on Intraglomerular Pressure in Hypertensive Patients
Brief Title: A Study to Evaluate the Effects of Manidipine Versus Amlodipine and the Combination of Manidipine Plus Delapril Versus Amlodipine Plus Delapril on Intraglomerular Pressure in Hypertensive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Principal Investigator, Roland E. Schmieder, Prof. Dr. med., University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-006350-10; MANTRA
Record Dates: First submitted 2008-02-24; First posted 2008-03-04 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Hypertension
Keywords: hypertension; intraglomerular pressure
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; manidipine; delapril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- amlodipine 10 mg (Active Comparator)
  Interventions: Drug: amlodipine 10 mg; Drug: amlodipine 5 mg + delapril 30 mg
- manidipine 20 mg (Active Comparator)
  Interventions: Drug: manidipine 20 mg; Drug: manidipine 10 mg + delapril 30 mg

INTERVENTIONS:
Drug: amlodipine 10 mg — amlodipine 10 mg once daily
  Arms: amlodipine 10 mg
Drug: manidipine 20 mg — manidipine 20 mg once daily
  Arms: manidipine 20 mg
Drug: amlodipine 5 mg + delapril 30 mg — amlodipine 5 mg + delapril 30 mg once daily
  Arms: amlodipine 10 mg
Drug: manidipine 10 mg + delapril 30 mg — manidipine 10 mg + delapril 30 mg once daily
  Arms: manidipine 20 mg

SUMMARY:
Eight-week multi-national, multicenter, randomized, double blind, active control, two arms, parallel groups study with a 4-week single drug treatment (manidipine or amlodipine) phase followed by a 4-week combination treatment (manidipine + delapril or amlodipine + delapril) phase.

DETAILED DESCRIPTION:
The aim of the current study is to assess the effect of a 4-week single drug treatment with manidipine or amlodipine and a 4-week combination treatment with manidipine plus delapril or amlodipine plus delapril on intraglomerular pressure in subjects with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients aged 18 years or older
* mild to moderate hypertension (systolic blood pressure > 139 mmHg or diastolic blood pressure > 89 mmHg)

Exclusion Criteria:

* secondary form of arterial hypertension
* severe hypertension (systolic blood pressure > 179 mmHg or diastolic blood pressure > 109 mmHg)
* pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
effect of manidipine 20 mg once daily compared to amlodipine 10 mg once daily on intraglomerular pressure | 4 weeks

SECONDARY OUTCOMES:
effects of combination of manidipine 10 mg plus delapril 30 mg once daily compared with once daily amlodipine 5 mg plus delapril 30 mg on intraglomerular pressure | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, Professor, Principal Investigator — University of Erlangen-Nürnberg
Locations (1):
- Clinical Research Center, Department of Nephrology and Hypertension, University of Erlangen-Nurnberg, Erlangen, Bavaria, Germany

REFERENCES:
- [Derived] Bosch AJ, Harazny JM, Kistner I, Friedrich S, Wojtkiewicz J, Schmieder RE. Retinal capillary rarefaction in patients with untreated mild-moderate hypertension. BMC Cardiovasc Disord. 2017 Dec 21;17(1):300. doi: 10.1186/s12872-017-0732-x. PMID 29268712